CLINICAL TRIAL: NCT01266408
Title: International Active Surveillance Study - Folate in Oral Contraceptives Utilization Study
Brief Title: INAS-FOCUS (International Active Surveillance Study - Folate in Oral Contraceptives Utilization Study)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2010_02; 15346 (Other: Bayer AG); EUPAS1597 (Registry Identifier: EUPAS Register)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Contraception
Keywords: Drospirenone; Dienogest; Metafolin; Folic acid; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DRSP/EE/metafolin: Women using oral contraceptives containing drospirenone, ethinylestradiol and metafolin
- Other OC users: Women using oral contraceptives containing other estrogen/progestogen combinations

SUMMARY:
The study compares the risks of short- and long-term use of contraceptives containing drospirenone (DRSP) or dienogest (DNG)/ethinylestradiol (EE) plus levomefolate calcium (metafolin) with the risks of short- and long-term use of other established oral contraceptives (OCs).

DETAILED DESCRIPTION:
New oral contraceptives (OCs) containing drospirenone (DRSP) or dienogest (DNG)/ethinylestradiol (EE) plus levomefolate calcium (metafolin) have been recently introduced and will be introduced in a number of countries in the near future. Although the safety of OCs has improved over the last 50 years with reductions in the estrogen and progestogen dose, special attention regarding oral contraceptive safety amongst women with risk factors for venous and arterial thromboembolism as well as cancer is necessary. Folic acid supplementation has been implicated in both the prevention and the promotion of several cancers, including colorectal cancer (CRC). Chronic folate deficiency seems to be associated with colorectal carcinogenesis, while high folic acid levels may have a tumor-promoting effect. On balance an oral contraceptive containing folate may be advantageous for several reasons. It may increase baseline folate levels with potential for protecting against some malignancies and concurrently decrease the risk of neural tube defects in women who become pregnant due to OC-failure, incorrect OC-use or after stopping the OC for a planned pregnancy. Although unexpected, it is unclear whether combined oral contraceptives plus metafolin in general and specifically DRSP/EE plus metafolin and DNG/EE plus metafolin will alter the risk profile of established oral contraceptives.

This study investigates the safety of these new oral contraceptives with regard to cardiovascular outcomes and colorectal cancer.

INAS-FOCUS is a prospective, controlled, non-interventional cohort study with three study arms: users of DRSP/EE/metafolin, users of DNG/EE/metafolin and users of OCs containing other estrogen/progestogen combinations. The users will be grouped to starters (first-ever users), switchers (women switching OC without a pill intake break) and restarters (women with a pill intake break). Users of an OC are accrued by a network of prescribing physicians. Baseline and follow-up information is collected via a self-administered questionnaire. Data analysis will be based on life-table methods comparing the cohorts.

Amendment, approved by the Safety Monitoring and Advisory Council on 13th May 2018:

During study recruitment, only one combined oral contraceptive was launched containing metafolin (DRSP/EE+) and the planned third cohort arm (users of DNG/EE+) was rendered obsolete.

In addition, early recruitment rates and exposure figures in INAS-FOCUS suggested that the study would be inadequately powered to accurately assess the risk of colorectal cancer at 15 years. Interim reports were presented to the Safety Monitoring and Advisory Council (SMAC) and in consultation with the funder, a decision made to discontinue INAS-FOCUS following analysis of cardiovascular events (Part 1 of study). The current protocol reflects the developments discussed above. The original three cohorts have been reduced to two (DRSP/EE+ and other OCs containing estrogen/progestogen) and Part II (long-term assessment of risk of colorectal cancer) has been removed from the protocol. Colorectal cancer outcomes will be analyzed as a secondary outcome for signal detection purposes only.

For historical accuracy and context, the introduction and background sections of the protocol have been left unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Women starting OC use ("starters")
* Women switching OC use without a pill intake break ("switchers")
* Women restarting OC use after a pill intake break ("restarters")
* Women willing to participate in the active surveillance

Exclusion Criteria:

* Long-term users
* Women who do not agree to participate
* Women with a language barrier

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women using oral contraceptives
Sampling Method: Non-Probability Sample
Enrollment: 82921 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Absolute risk of Venous Thromboembolic Events | Within 6 years
Absolute risk of Acute Myocardial Infarction | Within 6 years
Absolute risk of Cerebrovascular Accidents | Within 6 years

SECONDARY OUTCOMES:
Colorectal cancer | Within 6 years
Other cancer entities | Within 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Dinger, PhD, MD, Principal Investigator — Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany